CLINICAL TRIAL: NCT00822952
Title: Prostate Mechanical Imager (PMI) Clinical Bridging Study
Acronym: PMI
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers, The State University of New Jersey (Other); Mayo Clinic (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PMI-03; 5R44CA082620 (NIH)
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Prostatic Neoplasms; Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate an imaging capability Prostate Mechanical Imager (PMI), a PC-based device utilizing a transrectal probe with pressure sensor arrays and motion tracking system, aimed at providing composite elasticity images of the prostate.

DETAILED DESCRIPTION:
The clinical application of a Prostate Mechanical Imaging (PMI) technique for prostate assessment is examined in this study. PMI technology is based on the visualization of internal structures and dimensions of the prostate by measuring mechanical stress patterns on the gland surface with pressure sensor arrays. Temporal and spatial changes in the stress pattern provide information on the hardness of the prostate. Projected patient sample size for the study is 40 men over the age of 21. Patients will be selected for the study if both of the following criteria are met: (1) abnormal DRE findings; and (2) patients who are scheduled for a TRUS-guided prostate biopsy and/ or radical prostatectomy due to an abnormal DRE, and/or increased PSA, and/or other clinical indications.

The study is designed to assess the imaging capability of the PMI in three clinical sites, performed by four physicians. Each clinical investigator will perform PMI examination on 10 respective patients with DRE detected abnormality. Pathology data will be collected from TRUS-guided biopsy or radical prostatectomy and will be used as reference data in case there is a discrepancy between the DRE findings and PMI images. Study Hypothesis: Proportion of patients with PMI reconstructed image is anticipated to be consistent with the 84% imaging capability demonstrated in the previous clinical study conducted with the prior version of the PMI device.

ELIGIBILITY:
Inclusion Criteria:

* all racial and ethnic groups,
* males 21 years of age or older,
* able to withstand body positioning for the entire length of examination,
* presence of DRE detected abnormality,
* scheduled for TRUS-biopsy or surgical removal or prostate,
* able to comprehend, sign, and date the written informed consent form (ICF)

Exclusion Criteria:

* previous pelvic surgery,
* significant hip and / vertebral arthritis,
* rectal Crohn's disease,
* locally disseminated cancer of pelvic structure,
* anal fissure, anal fistula, infected anal fistula,
* anal cancer,
* rectal cancer,
* 1st, 2nd or 3rd degree hemorrhoids,
* pelvic irradiation,
* dehydrated impacted stool,
* no vulnerable patients such as students, nursing home residents, institutionalized patients, and those with psychological or physical incapacity will be included in the study

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male patients between over the age of 21 presenting to the participating clinical sites for urologic examination with the DRE detected prostate abnormality and scheduled for a TRUS-guided prostate biopsy and/ or radical prostatectomy due to an abnormal DRE, and/or increased PSA, and/or other clinical indications will be considered for inclusion. All ethnic and racial groups will be included.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Prostate Mechanical Imager provides reconstructed image of prostate | 1 Year

SECONDARY OUTCOMES:
Prostate Mechanical Imager recorded images of prostate are consistent with the abnormal digital rectal examination findings | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, Ph.D., D.Sc., Principal Investigator — Artann Laboratories
Locations (5):
- United States (5):
  - University of Minnesota/VA Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Urology Associates of Lancaster, Lancaster, Pennsylvania

REFERENCES:
- [Background] Weiss RE, Egorov V, Ayrapetyan S, Sarvazyan N, Sarvazyan A. Prostate mechanical imaging: a new method for prostate assessment. Urology. 2008 Mar;71(3):425-9. doi: 10.1016/j.urology.2007.11.021. PMID 18342178
- See also: Artann Laboratories — http://www.artannlabs.com